CLINICAL TRIAL: NCT04979819
Title: The Validity and Reliability of the Upper Extremity Exercise Testing (UULEX) in Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2021.770
Record Dates: First submitted 2021-07-27; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Validity and Reliability
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple Sclerosis (Experimental): Patients with multiple sclerosis will perform the UULEX and fill in the other mentioned parameters. Validity and reliability of the UULEX will be measured.
  Interventions: Other: Upper extremity endurance test (UULEX)

INTERVENTIONS:
Other: Upper extremity endurance test (UULEX) — Patients will lift 5 bars consecutively rhythmically until they feel fatigued. The bars will weigh 200 grs 500 gr 1kgs and 2 kgs respectively. The duration of the test will be measured to determine the endurance levels of the patients.

SUMMARY:
Multiple sclerosis negatively affects the endurance and functionality in the upper extremities. 20 female patients aged 18-70 years who were diagnosed with MS will be included in the study. Demographic, family, cigarette alcohol use, etc. information will be obtained from the patients and the study will begin. Timed 25-Step Walking Test, upper extremity endurance with UULEX, Hand-Shoulder and Arm Problems Questionnaire (DASH) and Nine-hole Board Test (DDTT) evaluation were performed on the patients. Manual muscle test for muscle strength, handheld dynamometer handheld Grip strength will be measured with a dynamometer and spasticity will be measured with the Ashworth scale. Depression status of the patients will be determined by the Beck depression scale, and the presence of dyspnea will be determined by the dyspnea scale.

The validity and reliability of the Unsupported Upper Extremity Exercise Test (UULEX) will be investigated with the obtained data. In order to give the most accurate result of the test in adults over 65 years of age, 3 repetitions will be performed with a resting period of half an hour.

Limitation of activities of daily living will be evaluated with MSQOL-54 specific to Multiple Sclerosis. Intraclass correlation coefficient (ICC) will be used to determine test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple scleroisis

Exclusion Criteria:

* Presence of extreme spasticity in the upper extremities that will prevent the performing of UULEX

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Upper extremity endurance testing | 1 day
  Upper extremity endurance testing

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided